CLINICAL TRIAL: NCT01031264
Title: Chronic Alcohol and Brain Stress Circuit Response
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Rajita Sinha, Professor, Yale University
Other Study IDs: 0706002821; R01AA013892 (NIH)
Record Dates: First submitted 2009-12-10; First posted 2009-12-14 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Stress; Alcoholism
Keywords: social drinkers
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Social drinkers

SUMMARY:
Alcoholism is among the top three causes of preventable death and disease in the US (Mokdad et al., 2004; Room et al., 2005). Stress plays an important role in the development of alcoholism and in high vulnerability to alcohol relapse. This study will provide a greater understanding of the mechanism by which stress and alcohol consumption interacts to influence development of compulsive alcohol seeking and vulnerability to stress-induced drinking, and the results will have significant implications for the development of new prevention and treatment interventions for alcoholism.

ELIGIBILITY:
Inclusion Criteria:

* ages 21-50

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: social drinkers
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2009-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Assess differences in reactivity to cue imagery | 2 years from start of study
  Physiological measures will be collected (heart rate, blood levels), self-reports of emotional states completed & alcohol taste task performed

CONTACTS AND LOCATIONS:
Overall Officials: Rajita Sinha, PhD, Principal Investigator — Yale University
Locations (1):
- Yale Stress Center, New Haven, Connecticut, United States